CLINICAL TRIAL: NCT00305383
Title: Analysis of Hepatitis C Viral Kinetics and Viramidine Pharmacokinetics Utilizing Two Treatment Regimens in Therapy-Naive Patients With Chronic Hepatitis C
Brief Title: Viral Kinetic Study With Viramidine in Therapy-Naive Patients With Chronic Hepatitis C
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Dose levels were determined to be subtherapeutic
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RNA003142-202
Record Dates: First submitted 2006-03-17; First posted 2006-03-21 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Hepatitis C, Chronic
Keywords: Viramidine; Peginterferon alfa-2b; Valeant; Hepatitis C; Rapid virologic response; HCV RNA
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — taribavirin; peginterferon alfa-2b

INTERVENTIONS:
Drug: Viramidine
Drug: Peginterferon alfa-2b

SUMMARY:
The purpose of this study is to examine the rapid virologic response (RVR) at combination therapy (CT) Week 4 between groups receiving a standard combination peginterferon alfa-2b/viramidine dosing regimen versus a cohort that receives 4 weeks of viramidine monotherapy prior to the start of peginterferon alfa-2b/viramidine combination therapy.

DETAILED DESCRIPTION:
This Phase 2b multicenter study, which is being conducted solely in the United States, consists of a randomized, double-blind, monotherapy period, where patients will receive either viramidine or placebo for 4 weeks. After the monotherapy period, all patients will receive viramidine plus peginterferon alfa-2b combination therapy for 48 weeks in an open-label fashion and will then participate in a 24-week follow-up period after completion of combination therapy. The RVR at CT Week 4 between groups receiving a standard combination peginterferon alfa-2b/viramidine dosing regimen versus a cohort that receives 4 weeks of viramidine monotherapy prior to the start of peginterferon alfa-2b/viramidine combination therapy will be examined. The differences in virological response during treatment and end of follow-up between African-Americans and Caucasians (non-Hispanics), as well as a correlation between duration of viral negativity (DVN) and sustained virologic response (SVR) based on race and dosing regimen, will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naive, genotype 1 only, compensated, chronic hepatitis C infected Caucasian or African-American patients
* Body weight greater than 61 kg and not more than 87.3 kg
* HCV RNA greater than 2 million copies/mL
* Elevated measured or historical alanine aminotransferase
* Hemoglobin at least 12.0 g/dL for females and at least 13.0 g/dL for males
* Calculated creatinine clearance greater than 70 mL/min

Exclusion Criteria:

* Cirrhosis of the liver
* Alanine aminotransferase greater than 3 times the upper limit of normal
* Severe neuropsychiatric disorders
* History or clinical manifestations of significant metabolic, hematological, pulmonary, ischemic, or unstable heart disease, gastrointestinal, neurological, renal, urological, endocrine, ophthalmologic disorders including severe retinopathy, or immune mediated disease
* Other co-morbid chronic viral infections including hepatitis B and the human immunodeficiency virus (HIV)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-11; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Efficacy: The proportion of patients with hepatitis C virus (HCV) RNA undetectable or with at least a 2-log drop from baseline at CT Week 4 in the viramidine pre-load group versus the viramidine standard dosing group.
Safety: Evaluation of adverse events (AEs).
Safety: Physical exams
Safety: Vital signs
Safety: Laboratory tests

SECONDARY OUTCOMES:
Efficacy: HCV RNA Response at CT Week 12, 24, end of treatment and at follow-up Week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph T. Doyle, Study Director — Bausch Health Americas, Inc.
Locations (11):
- United States (11):
  - University of Southern California -- Keck School of Medicine, Los Angeles, California
  - San Mateo Medical Center, San Mateo, California
  - Bach and Godofsky, Bradenton, Florida
  - University of Miami -- Center for Liver Diseases, Miami, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Maryland Digestive Disease Research, Laurel, Maryland
  - Atlantic Gastroenterology Associates, Egg Harbor, New Jersey
  - Liver Center of Long Island, Plainview, New York
  - Thomas Jefferson University -- Gastroenterology and Hepatology, Philadelphia, Pennsylvania
  - Mountain West Gastroenterology -- Research Office, Salt Lake City, Utah
  - Metropolitan Research -- Georgetown Medical Center, Fairfax, Virginia